CLINICAL TRIAL: NCT05452707
Title: Task-oriented Arm/Hand Skill Rehabilitation and Therapy Dose Dimensions in Subacute Spinal Cord Injury Rehabilitation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hasselt University (Other)
Collaborators: Adelante Zorggroep (Unknown); Universitaire Ziekenhuizen KU Leuven (Other); University Ghent (Other)
Responsible Party: Principal Investigator, Annemie Spooren, Principal Investigator, Hasselt University
Other Study IDs: NB1
Record Dates: First submitted 2022-04-06; First posted 2022-07-11 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-04

CONDITIONS: Spinal Cord Injuries
Keywords: Spinal cord rehabilitation; Therapy content in arm/hand skill training; Therapy dose in spinal cord rehabilitation
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Observation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients: Patients will be observed during their active training sessions.
  Patients will be asked questions about:
  * fatigue
  * physical fatigue
  * pain
  * the difficulty of the session
  * motivation
  Interventions: Other: Observation and questionnaire of active therapy
- Therapists: Therapists will be asked questions about the observed training sessions of the patients. The questions will be about:
  * Estimation of active training time
  * Estimation of patient's fatigue
  * Estimation of the patient's perceived difficulty of the session
  * Estimation of the patient's perceived physical fatigue of the session
  * Estimation of the patient's perceived motivation for the session
  Interventions: Other: Observation and questionnaire of active therapy

INTERVENTIONS:
Other: Observation and questionnaire of active therapy — There will be an observation of the usual care; no intervention will be added.

SUMMARY:
The study is a multicenter longitudinal observational study. The therapy content and the therapy dosage of arm/skill training for patients with cervical spinal cord injury (SCI) will be observed for the primary objective. The aim is to get insight into the current therapy content and the current therapy dosage in arm/hand skill training, with the overall aim to optimize the arm/hand skill training. For the secondary objective, in addition to the patients with cervical SCI also, patients with paraplegia as a result of SCI are included. The aim is to assess the difference between the patient's perceived dose and the therapist's estimation of the therapy dose. This will give insight into the patient's and therapist's views on therapy dose; this information will contribute to optimizing therapy dose in exercise therapy in SCI. The third aim is a pilot study to explore the usability of evening reports in SCI rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Primary objective

  1. Have sustained a traumatic or non-traumatic SCI between C1 and T1.
  2. Have an AIS A, B, C or D
  3. Are older than 16 years
  4. Being able to follow standard arm/hand skill training.
  5. Patients in the subacute phase (4-30 weeks post-injury)
  6. Receiving usual care
  7. Able to understand the purpose of the study (understanding Dutch, English, French and German).
* Secondary objective

Add patients with:

1. Persons with SCI (C1-S4)
2. having an AIS A, B, C, D;
3. Are older than 16 years;
4. Patients in the subacute phase (4-30 weeks post-injury)
5. receiving standard care or more intensive care as defined by the SCI-MT trial - Therapists Physiotherapists, occupational therapists and sports therapists with at least two years of experience in SCI rehabilitation

Exclusion Criteria:

1. have any significant medical or physical condition (including pregnancy) or psychiatric illness that could prevent the person from participating in the study
2. are unable/unwilling to provide informed consent.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients during the subacute phase (0-12 months post-injury) of a spinal cord injury.
  Therapists who give active training to patients in the subacute phase (0-12 months post-injury) of a spinal cord injury.
Sampling Method: Non-Probability Sample
Enrollment: 47 (Estimated)
Dates: Start 2022-07-11 (Actual); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
Task-oriented and therapy dose dimensions and the change in time of these components in arm/hand skill training in usual care in cervical SCI during subacute rehabilitation | Patients will be observed for three weeks between 4 and 20 weeks post-injury. There will be three random days of observations. Data will be collected from every therapy session with at least 50% arm/hand skill training
  * An observer reports the therapy content (endurance training, strength training and skill training) on a data report
  * Active training time is measured with accelerometers on both wrists
  * An observer with a hand counter measures movement repetitions
  * The prescribed, planned and given therapy hours are reported on a data form

SECONDARY OUTCOMES:
Perceived dose in spinal cord injury in the subacute rehabilitation | Patients will be observed for three weeks between 4 and 20 weeks post-injury. There will be three random days of observations. Data will be collected before and after every active therapy session.
  Patients and therapists answers questions before and after the sessions
  Patients get questions on:
  * Fatigue
  * Pain
  * Difficulty
  * Physical fatigue
  * Motivation
  Therapists get questions on:
  * Estimation of active training time
  * Estimation of patient's fatigue
  * Estimation of the patient's perceived difficulty of the session
  * Estimation of the patient's perceived physical fatigue of the session
  * Estimation of the patient's perceived motivation of the session

OTHER OUTCOMES:
Pilot study: usability of evening reports in rehabilitation of SCI. | Patients will be observed for three weeks between 4 and 20 weeks post-injury. There will be three random days of observations. Data will be collected in the evening after the active therapy session.
  Patients get questions on a evening report the themes are:
  * Pain
  * Fatigue
  * Motivation
  * Satisfaction
  * Acceptance
  * General mood
  Patients get questions on a evening report the themes are:
  * Pain
  * Fatigue
  * Motivation
  * Satisfaction
  * Acceptance
  * General mood

CONTACTS AND LOCATIONS:
Overall Officials: Annemie Spooren, Prof.Dr., Principal Investigator — UHasselt
Locations (3):
- Belgium (2):
  - UZ Gent, Ghent
  - UZ Leuven - Campus Pellenberg, Leuven
- Zorggroep Adelante, Hoensbroek, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided